CLINICAL TRIAL: NCT06324968
Title: Ro60 Expression in Macrophages in Patients with Primary Sjogren's Syndrome
Brief Title: Ro60 Expression in Macrophages in Sjogren's Disease
Acronym: RoMioSS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-AOIP-01
Record Dates: First submitted 2023-12-19; First posted 2024-03-22 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Sjogren's Syndrome
Keywords: Sjogren's Syndrome; cardiovascular risk; Ro60; protein; connective tissue disorder
MeSH Terms: conditions — Sjogren's Syndrome; Connective Tissue Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sjögren's disease (Experimental): SSp patients followed by the Internal Medicine Department of Nice University Hospital will be offered participation in this study as part of their usual follow-up.
  Interventions: Diagnostic Test: Positive serology for anti-SSA
- Control (No Intervention): Control subjects will be recruited from the nursing staff of Nice University Hospital on a voluntary basis.

INTERVENTIONS:
Diagnostic Test: Positive serology for anti-SSA — Blood sample which detect serology for anti-SSA.
  Arms: Sjögren's disease

SUMMARY:
Context: The Ro60 protein associates with YRNAs (or RNYs) to form the RoRNP complex, which regulates RNA surveillance and maturation. It is hypothesized that its impairment by nuclear penetration of the anti-Ro60 autoantibodies, would deregulate the anti-inflammatory response in monocytes/macrophages (Mo/Mp) in patients with Sjögren's disease (SD).

ELIGIBILITY:
Inclusion Criteria:

* Patients with SSp Subjects aged between 18 and 75, without chronic disease; Subject meeting the classification criteria for SSp; Subject with positive anti-SSA serology; French-speaking subject able to give written consent; Subject affiliated to the Sécurité Sociale or an equivalent scheme; Subject willing to have blood samples taken;
* Control subjects Subjects aged between 18 and 75, without chronic disease and not meeting SSp classification criteria; Subject who understands and speaks French and is able to give written consent; Subject affiliated to the French Social Security system or an equivalent scheme; Subject willing to have blood taken;

Exclusion Criteria:

* Subject receiving current anti-inflammatory treatment (e.g. corticosteroid therapy, non-steroidal anti-inflammatory drugs) or a regimen of more than 1 month within the last 3 months;
* Subject undergoing biotherapy or cytoreductive treatment;
* Subjects with positive serologies for human immunodeficiency virus (HIV), viral hepatitis B virus (HBV) and viral hepatitis C virus (HCV) in the 3 months preceding the inclusion visit;
* Protected persons as defined in articles of the French Public Health Code.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2025-05-09 (Estimated)

PRIMARY OUTCOMES:
SSA/Ro60 interactions | 1 year
  To evaluate whether the presence of anti-Ro60 autoantibodies causes the loss of Ro60 binding activity to genomic DNA and the TREX protein complex in PBMC.
  Measure the presence of anti-Ro60 autoantibodies in blood.

SECONDARY OUTCOMES:
The molecular and functional impact : inflammatory cytokine and chemokine profiles | 1 year
  To explore the molecular and functional impact of the anti-Ro60 autoantibodies in Mo/Ma to gain insights into the pathological relevance by evaluating inflammatory cytokine and chemokine profiles with using the ELISA (Enzyme Linked Immuno Sorbent Assay) technique.
The molecular and functional impact : cell apoptosis/survival and cellular polarization | 1 year
  To explore the molecular and functional impact of the anti-Ro60 autoantibodies in Mo/Ma to gain insights into the pathological relevance by assessing cell apoptosis/survival and cellular polarization with flow-cytometry analysis.
The molecular and functional impact : clinical and biochemical phenotypes of CD14+ monocytes/macrophages | 1 year
  To explore the molecular and functional impact of the anti-Ro60 autoantibodies in Mo/Ma to gain insights into the pathological relevance by comparing clinical and biochemical phenotypes of CD14+ monocytes/macrophages by labeling with Monoclonal Antibodies then count the number of cells.

CONTACTS AND LOCATIONS:
Overall Officials: Nihal MARTIS, MD, MSc, Principal Investigator — CHU NICE
Locations (1):
- CHU Nice, Nice, Alpes-Mritimes, France

IPD SHARING:
Plan to Share IPD: No